CLINICAL TRIAL: NCT00694252
Title: A Pilot Feasibility Study to Evaluate the Efficacy of Lapatinib in Eliminating Cytokeratin-positive Tumour Cells Circulating in the Blood of Women With Breast Cancer
Brief Title: Lapatinib and Circulating Tumor Cells in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, Prof. V.Georgoulias, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.15
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Tykerb; CTCs
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Lapatinib
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — Patients will receive lapatinib monotherapy 1500 mg/day for a period of at least one month depending on their response and the clinical status of their disease.
  Other Names: Tykerb; Tyverb; GW572016

SUMMARY:
This study will evaluate the efficacy of lapatinib in eradicating chemo- resistant tumour cells circulating in the blood of patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is considered a systemic disease since early tumour cell dissemination may occur even in patients with small tumours; several investigators using immunocytochemistry or real time PCR (RT-PCR) have shown that cytokeratin-positive epithelial cells could be identified in the bone marrow aspirates or the peripheral blood of otherwise metastases-free patients with stage I and II breast cancer. The clinical importance of the immunocytochemical detection of occult tumour cells in the bone marrow has been confirmed in many prospective studies to represent an independent predictive and prognostic factor for distant relapse and reduced survival.

Patients with metastatic breast cancer who have persistent detection of tumour cells in the peripheral blood (≥5 cells/7.5 ml) despite at least one line of chemotherapy will receive lapatinib for a minimum of one month unless disease progression occurs at an earlier time point.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Histologically or cytologically confirmed breast cancer
* Metastatic breast cancer (stage IIIB and IV). EGFR and/or HER-2 expression on the primary tumor is not mandatory.
* Patients should have received at least one course of standard systemic chemotherapy for their metastatic disease. Prior hormonal therapy is allowed.
* Patients should have achieved objective response (CR or PR) or stable disease to previous first or second line treatment.
* There should be at least one month between the end of chemotherapy treatment and trial entry. In case of prior Herceptin administration, 3 months are required to have elapsed before study entry.
* Detection of ≥5 cells/7.5ml of peripheral blood detected by Cell Search System despite the previous administration of chemotherapy and/or hormonal therapy.
* HER-2 expression on CTCs.
* Age 18 years and over
* Adequate Haematological function, Absolute neutrophil count ≥1.5 x 109/L, Platelet count ≥100 x 109/L and Haemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level)
* Adequate Liver Function, total bilirubin <1.5 x upper limit of normal, AST and ALT <2.5 x upper limit of normal in patients without liver metastases and <5 x upper limit of normal in patients with liver metastases
* Adequate Renal function, Serum creatinine ≤1.25 x upper limit of normal or calculated creatinine clearance ≥50 mL/min
* LVEF within institutional normal range
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Any concurrent systemic treatment for breast cancer (including chemotherapy, radiotherapy, hormonotherapy, monoclonal antibodies)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity greater than Grade 2 (NCI- CTCAE) from previous anticancer therapy (except alopecia)
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Pregnancy or breast feeding (women of child-bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment
* Known hypersensitivity to drugs chemically related to lapatinib
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of lapatinib by quantitative analysis of circulating tumour cells in the blood.The efficacy will be measured before, during and after the completion of treatment | 2 months

SECONDARY OUTCOMES:
Correlation of the levels of CTCs with the PFS of the patients | 1 year
Assessment of the safety of lapatinib administration in this patient population. | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Aggelaki, MD, Principal Investigator — University Hospital of Crete
Locations (1):
- University Hospital of Crete, Heraklion, Greece

REFERENCES:
- [Derived] Agelaki S, Kalykaki A, Markomanolaki H, Papadaki MA, Kallergi G, Hatzidaki D, Kalbakis K, Mavroudis D, Georgoulias V. Efficacy of Lapatinib in Therapy-Resistant HER2-Positive Circulating Tumor Cells in Metastatic Breast Cancer. PLoS One. 2015 Jun 17;10(6):e0123683. doi: 10.1371/journal.pone.0123683. eCollection 2015. PMID 26083256